CLINICAL TRIAL: NCT01215227
Title: A Phase 3, 40-Week, Active-Controlled, Double-Blind, Double-Dummy Extension Study of Preladenant in Subjects With Moderate to Severe Parkinson's Disease (Phase 3, Protocol No. P06153)
Brief Title: An Active-Controlled Extension Study to NCT01155466 [P04938] and NCT01227265 [P07037] (P06153)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P06153; 2009-015162-57 (EudraCT Number)
Record Dates: First submitted 2010-10-04; First posted 2010-10-06 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-10

CONDITIONS: Parkinson Disease; Idiopathic Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — 2-(2-furanyl)-7-(2-(4-(4-(2-methoxyethoxy)phenyl)-1-piperazinyl)ethyl)-7H-pyrazolo(4,3-e)(1,2,4)triazolo(1,5-c)pyrimidine-5-amine; rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Preladenant 2 mg (Experimental): Participants who received preladenant 2 mg in parent study NCT01155466 or NCT01227265 will continue to receive preladenant 2 mg in this extension study. Participants will receive preladenant 2 mg taken orally twice daily (BID): one tablet plus placebo capsule to rasagiline in the morning, and one tablet in the evening, for 40 weeks.
  Interventions: Drug: Preladenant; Drug: Placebo to rasagiline
- Preladenant 5 mg (Experimental): Participants who received preladenant 5 mg in parent study NCT01155466 or NCT01227265 will continue to receive preladenant 5 mg in this extension study. Participants will receive preladenant 5 mg taken orally BID: one tablet plus placebo capsule to rasagiline in the morning, and one tablet in the evening, for 40 weeks.
  Interventions: Drug: Preladenant; Drug: Placebo to rasagiline
- Preladenant 5 mg (on placebo in parent study) (Experimental): Participants who received placebo to preladenant tablet in parent study NCT01155466 or NCT01227265 will receive preladenant 5 mg in this extension study. Participants will receive preladenant 5 mg taken orally BID: one tablet plus placebo capsule to rasagiline in the morning, and one tablet in the evening, for 40 weeks.
  Interventions: Drug: Preladenant; Drug: Placebo to rasagiline
- Preladenant 10 mg (Experimental): Participants who received preladenant 10 mg in parent study NCT01155466 or NCT01227265 will continue to receive preladenant 10 mg in this extension study. Participants will receive preladenant 10 mg taken orally BID: one tablet plus placebo capsule to rasagiline in the morning, and one tablet in the evening, for 40 weeks.
  Interventions: Drug: Preladenant
- Rasagiline 1 mg (Active Comparator): Participants who received rasagiline 1 mg in parent study NCT01155466 or NCT01227265 will continue to receive rasagiline 1 mg in this extension study. Participants will receive rasagiline 1 mg capsule once a day: one capsule plus placebo tablet to preladenant in the morning, and one placebo tablet to preladenant in the evening, for 40 weeks.
  Interventions: Drug: Rasagiline; Drug: Placebo to preladenant
- Rasagiline 1 mg (on placebo in parent study) (Active Comparator): Participants who received placebo to rasagiline capsule in parent study NCT01155466 or NCT01227265 will receive rasagiline 1 mg in this extension study. Participants will receive rasagiline 1 mg capsule once a day: one capsule plus placebo tablet to preladenant in the morning, and one placebo tablet to preladenant in the evening, for 40 weeks.
  Interventions: Drug: Rasagiline; Drug: Placebo to preladenant

INTERVENTIONS:
Drug: Preladenant — Daily for 40 weeks: 2, 5, or 10 mg preladenant tablet each morning; 2, 5, or 10 mg preladenant tablet each evening (approximately 8 hours after the morning dose)
  Other Names: SCH 420814
  Arms: Preladenant 10 mg; Preladenant 2 mg; Preladenant 5 mg; Preladenant 5 mg (on placebo in parent study)
Drug: Rasagiline — Daily for 40 weeks: 1 mg rasagiline capsule each morning
  Other Names: Azilect®
  Arms: Rasagiline 1 mg; Rasagiline 1 mg (on placebo in parent study)
Drug: Placebo to preladenant — Placebo to match preladenant given daily for 40 weeks: placebo tablet each morning; placebo tablet each evening (approximately 8 hours after the morning dose)
  Arms: Rasagiline 1 mg; Rasagiline 1 mg (on placebo in parent study)
Drug: Placebo to rasagiline — Placebo to match rasagiline given daily for 40 weeks: placebo capsule each morning
  Arms: Preladenant 2 mg; Preladenant 5 mg; Preladenant 5 mg (on placebo in parent study)

SUMMARY:
The primary purpose of this extension study is to assess the long-term safety and tolerability of preladenant in participants from parent studies NCT01155466 [P04938] and NCT01227265 [P07037] with moderate to severe Parkinson's Disease (PD). The study will also characterize the long-term efficacy of preladenant in participants with PD.

Participants will continue to receive their stable regimen of levodopa (L-dopa) plus any adjunct medications during the study as prescribed by their physician. Several classes of adjunct medications may be used, including Amantadine, anticholinergics, dopa decarboxylase inhibitors, and dopamine agonists.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have completed the 12-week treatment period of the parent trial, P04938 or P07037.
* Participants must be willing and able to provide written informed consent for P06153.
* Participants must be able to adhere to dose and visit schedules.
* Participants must be taking L-dopa.
* Participants may be taking additional adjunct PD medications (e.g., dopamine agonists, entacapone).
* Each participant must have results of clinical laboratory tests (hematology, blood chemistries, and urinalysis) within normal limits or clinically acceptable to the investigator as evidenced by the last available test results from the parent study (P04938 or P07037), and no results fall within the parameters for exclusion described below in the exclusion criterion for liver-related findings.
* There has been no change in, or there has been no finding to warrant checking, serology status (for cytomegalovirus [CMV], Epstein-Barr virus [EBV], and Hepatitis B, C, and E).
* Each participant must have results of a physical examination within normal limits, including blood pressure, within normal limits or clinically acceptable limits to the investigator, and not within the parameters for exclusion described below in the exclusion criterion for blood pressure.
* All participants who are sexually active or plan to be sexually active agree to use a highly effective method of birth control while the participant is in the study and for 2 weeks after the last dose of study drug. A male participant must not donate sperm within 2 weeks after the last dose of study drug.

Exclusion Criteria:

* Any participant who discontinued from P04938 or P07037 for any reason.
* Any participant with a severe or ongoing unstable medical condition (e.g., any form of clinically significant cardiac disease, symptomatic orthostatic hypotension, seizures, or alcohol/drug dependence).
* Any participant with a history of poorly controlled diabetes (e.g., hemoglobin A1c > 8.5) or significantly abnormal renal function (e.g., creatinine > 2.0 mg/dL) in the opinion of the investigator.
* As a continuation of the liver-related withdrawal criteria from the parent studies (P04938 and P07037), any participant with elevated values for alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin (T BIL), as evidenced by the most recent chemistry panel results in the parent study, meeting any one of the following criteria:
* ALT or AST > 8 x upper limit of normal (ULN).
* ALT or AST > 5 x ULN for more than 2 weeks.
* ALT or AST > 3 x ULN and (T-BIL > 2 x ULN or international normalized ratio [INR] > 1.5 that is not due to anti-coagulation) at the same visit.
* ALT or AST > 3 x ULN with the appearance of worsening fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (> 5%).
* As a continuation of the blood pressure (BP) withdrawal criteria from the parent study (P04938 or P07037), any participant meeting the following criteria for the second of two consecutive visits separated by 7 days (i.e., the participant met one of the BP criteria once already, 7 days before the P06153 screening visit):
* Systolic BP ≥ 180 mm Hg or diastolic BP ≥ 105 mm Hg, or
* An elevation from baseline BP in the parent study (P04938 or P07037) of systolic BP >= 40 mm Hg or diastolic BP ≥ 20 mm Hg.
* A participant must not have a history within the past 5 years of a primary or recurrent malignant disease with the exception of adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or in situ prostate cancer with a normal prostate-specific antigen (PSA) post resection.
* Any participant with an average daily consumption of more than three 4-ounce glasses (118 mL) of wine or the equivalent.
* A participant must not have received certain prespecified medications or ingested high tyramine-containing aged cheeses (e.g., Stilton) for a prespecified time window before the trial, during the trial, and for 2 weeks after the trial.
* Any participant with allergy/sensitivity to the investigational products or their excipients.
* Any female participant breast feeding or considering breast feeding.
* Any female participant pregnant or intending to become pregnant.
* Any participant with any clinically significant condition or situation, other than the condition being studied that, in the opinion of the investigator, would interfere with the trial evaluations or optimal participation in the trial.
* Any participant with a member or a family member of the personnel of the investigational or sponsor staff directly involved with this trial.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 839 (Actual)
Dates: Start 2010-11-18 (Actual); Primary Completion 2013-07-16 (Actual); Study Completion 2013-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Preladenant 2 mg: Participants who received preladenant 2 mg in parent study NCT01155466 or NCT01227265 continued to receive preladenant 2 mg in this extension study. Participants received preladenant 2 mg taken orally twice daily (BID): one tablet plus placebo capsule to rasagiline in the morning, and one tablet in the evening, for 40 weeks.
- Preladenant 5 mg: Participant who received preladenant 5 mg in parent study NCT01155466 or NCT01227265 continued to receive preladenant 5 mg in this extension study. Participants received preladenant 5 mg taken orally BID: one tablet plus placebo capsule to rasagiline in the morning, and one tablet in the evening, for 40 weeks.
- Preladenant 5 mg (on Placebo in Parent Study): Participants who received placebo to preladenant tablet in parent study NCT01155466 or NCT01227265 received preladenant 5 mg in this extension study. Participants received preladenant 5 mg taken orally BID: one tablet plus placebo capsule to rasagiline in the morning, and one tablet in the evening, for 40 weeks.
- Preladenant 10 mg: Participants who received preladenant 10 mg in parent study NCT01155466 or NCT01227265 continued to receive preladenant 10 mg in this extension study. Participants received preladenant 10 mg taken orally BID: one tablet plus placebo capsule to rasagiline in the morning, and one tablet in the evening, for 40 weeks.
- Rasagiline 1 mg: Participants who received rasagiline 1 mg in parent study NCT01155466 or NCT01227265 continued to receive rasagiline 1 mg in this extension study. Participants received rasagiline 1 mg capsule once a day: one capsule plus placebo tablet to preladenant in the morning, and one placebo tablet to preladenant in the evening, for 40 weeks.
- Rasagiline 1 mg (on Placebo in Parent Study): Participants who received placebo to rasagiline capsule in parent study NCT01155466 or NCT01227265 received rasagiline 1 mg in this extension study. Participants received rasagiline 1 mg capsule once a day: one capsule plus placebo tablet to preladenant in the morning, and one placebo tablet to preladenant in the evening, for 40 weeks.
Period: Overall Study
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 5 mg (on Placebo in Parent Study) | Preladenant 10 mg | Rasagiline 1 mg | Rasagiline 1 mg (on Placebo in Parent Study)
Started | 218 | 215 | 107 | 97 | 93 | 109
Treated | 218 | 215 | 106 | 96 | 93 | 108
Completed | 97 | 96 | 50 | 48 | 45 | 51
Not Completed | 121 | 119 | 57 | 49 | 48 | 58
Not completed — Adverse Event | 11 | 11 | 4 | 8 | 7 | 6
Not completed — Treatment Failure | 8 | 4 | 1 | 5 | 1 | 1
Not completed — Lost to Follow-up | 1 | 4 | 1 | 1 | 1 | 2
Not completed — Subject Withdrew Consent | 16 | 20 | 7 | 10 | 11 | 8
Not completed — Non-Compliance With Protocol | 2 | 6 | 1 | 0 | 0 | 0
Not completed — Administrative | 83 | 73 | 42 | 24 | 28 | 40
Not completed — Missing Status | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Randomized but not treated | 0 | 0 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All Participants as Treated: All participants who received at least one dose of study drug in Extension Study P06153. Data were not reported for 3 participants who were randomized but not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 5 mg (on Placebo in Parent Study) | Preladenant 10 mg | Rasagiline 1 mg | Rasagiline 1 mg (on Placebo in Parent Study) | Total
Number analyzed (Participants) | 218 | 215 | 106 | 96 | 93 | 108 | 836
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.4 (8.5) | 63.0 (8.7) | 64.4 (8.7) | 63.9 (8.0) | 63.8 (9.9) | 63.9 (7.8) | 63.3 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 100 | 55 | 40 | 37 | 41 | 341
  Male | 150 | 115 | 51 | 56 | 56 | 67 | 495

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Systolic Blood Pressure ≥180 mmHg
Description: The percentage of participants with Systolic Blood Pressure ≥180 mm Hg was reported. On Day 1 and Early Termination, blood pressure was measured as follows: Participant lay supine for 5 minutes, then had blood pressure taken; then stood for 3 minutes and had blood pressure taken; then rested for 10 minutes, at which time the process was repeated twice (ie, three rounds total). For all other blood pressure measurements, the procedure needed only to be done once (ie, one round).
Time Frame: Up to 42 weeks
Population: All Participants as Treated (APaT) population, which consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 5 mg (on Placebo in Parent Study) | Preladenant 10 mg | Rasagiline 1 mg | Rasagiline 1 mg (on Placebo in Parent Study)
Number analyzed (Participants) | 218 | 215 | 106 | 96 | 93 | 108
Percentage of participants | 1.4 | 0.0 | 0.9 | 1.0 | 0.0 | 0.9

2. Primary Outcome: Percentage of Participants With Diastolic Blood Pressure ≥105 mmHg
Description: The percentage of participants with Diastolic Blood Pressure ≥105 mmHg was reported. On Day 1 and Early Termination, blood pressure was measured as follows: Participant lay supine for 5 minutes, then had blood pressure taken; then stood for 3 minutes and had blood pressure taken; then rested for 10 minutes, at which time the process was repeated twice (ie, three rounds total). For all other blood pressure measurements, the procedure needed only to be done once (ie, one round).
Time Frame: Up to 42 weeks
Population: APaT population, which consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 5 mg (on Placebo in Parent Study) | Preladenant 10 mg | Rasagiline 1 mg | Rasagiline 1 mg (on Placebo in Parent Study)
Number analyzed (Participants) | 218 | 215 | 106 | 96 | 93 | 108
Percentage of participants | 5.0 | 4.2 | 5.7 | 5.2 | 7.5 | 8.3

3. Primary Outcome: Percentage of Participants With Alanine Aminotransferase (ALT) ≥3 Times Upper Limit of Normal and ≥10% Increase From Baseline
Description: The number of participants with ALT ≥3 times the upper limit of normal and a ≥10% increase was reported. Laboratory safety blood work was collected from participants at Week 4, Week 6, and Week 8 visits.
Time Frame: Up to 42 weeks
Population: APaT population, which consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 5 mg (on Placebo in Parent Study) | Preladenant 10 mg | Rasagiline 1 mg | Rasagiline 1 mg (on Placebo in Parent Study)
Number analyzed (Participants) | 218 | 215 | 106 | 96 | 93 | 108
Percentage of participants | 1.4 | 0.5 | 0.0 | 1.0 | 0.0 | 1.9

4. Primary Outcome: Percentage of Participants With Aspartate Aminotransferase (AST) ≥3 Times Upper Limit of Normal and ≥10% Increase From Baseline
Description: The number of participants with AST ≥3 times the upper limit of normal and a ≥10% increase was reported. Laboratory safety blood work was collected from participants at Week 4, Week 6, and Week 8 visits.
Time Frame: Up to 42 weeks
Population: APaT population, which consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 5 mg (on Placebo in Parent Study) | Preladenant 10 mg | Rasagiline 1 mg | Rasagiline 1 mg (on Placebo in Parent Study)
Number analyzed (Participants) | 218 | 215 | 106 | 96 | 93 | 108
Percentage of participants | 1.4 | 0.5 | 0.0 | 2.1 | 1.1 | 2.8

5. Primary Outcome: Percentage of Participants With Suicidality
Description: The number of participants with suicidality using the Columbia - Suicide Severity Rating Scale (C-SSRS) was reported. The C-SSR was used in this study only for the purpose of safety monitoring by measuring the incidence of different types of suicidality categories during treatment. The assessment was done by the nature of the responses, not by a numbered scale. Participants who reported at least one occurrence of suicidal behavior or suicidal ideation were counted as having experienced suicidality. Suicidal behavior included suicide attempt, aborted attempt, interrupted attempt, or preparatory behavior. Suicidal ideation included a wish to die or active suicidal thought with or without method, intent or plan.
Time Frame: Up to 42 weeks
Population: APaT population, which consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 5 mg (on Placebo in Parent Study) | Preladenant 10 mg | Rasagiline 1 mg | Rasagiline 1 mg (on Placebo in Parent Study)
Number analyzed (Participants) | 218 | 215 | 106 | 96 | 93 | 108
Percentage of participants | 4.1 | 5.6 | 0.0 | 4.2 | 2.2 | 2.8

6. Primary Outcome: Percentage Change From Baseline in Total Epworth Sleepiness Scale (ESS) Score at Week 40
Description: The ESS is a self-administered questionnaire providing a measure of a person's general level of daytime sleepiness, or their average sleep propensity in daily life. The scale consists of 8 situations in which the participant rates their tendency to become sleepy on a scale of 0=no chance of dozing to 3=high chance of dozing. The overall score is the sum of the scores for the 8 situations for a minimum of 0 and a maximum of 24 with a higher score indicating greater sleepiness.
Time Frame: Baseline and Week 40
Population: Participants in the Full Analysis Set (FAS) population (all randomized participants who received at least one dose of study drug) that had a baseline value and data at Week 40 for Total ESS Score
Measure: Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 5 mg (on Placebo in Parent Study) | Preladenant 10 mg | Rasagiline 1 mg | Rasagiline 1 mg (on Placebo in Parent Study)
Number analyzed (Participants) | 90 | 88 | 47 | 49 | 48 | 49
Percentage change | 15.5 (3.4) [-15.0 to 46.2] | 24.0 (3.9) [7.8 to 40.3] | 22.5 [-9.5 to 54.5] | 13.2 [-5.9 to 32.4] | 8.3 [-6.8 to 23.4] | 16.3 [-3.3 to 35.9]

ADVERSE EVENTS:
Time Frame: Up to 42 weeks
Description: APaT population, which consisted of all participants who received at least one dose of study drug.
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 5 mg (on Placebo in Parent Study) | Preladenant 10 mg | Rasagiline 1 mg | Rasagiline 1 mg (on Placebo in Parent Study)
Serious Adverse Events (participants affected / at risk) | 11/218 | 15/215 | 6/106 | 12/96 | 5/93 | 4/108
Other Adverse Events (participants affected / at risk) | 64/218 | 71/215 | 30/106 | 35/96 | 25/93 | 38/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preladenant 2 mg (N=218) | Preladenant 5 mg (N=215) | Preladenant 5 mg (on Placebo in Parent Study) (N=106) | Preladenant 10 mg (N=96) | Rasagiline 1 mg (N=93) | Rasagiline 1 mg (on Placebo in Parent Study) (N=108)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERTENSIVE CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SICK SINUS SYNDROME (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
HIATUS HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ILEUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VOLVULUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST DISCOMFORT (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALAISE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHOPNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENCEPHALITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NOSOCOMIAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OROPHARYNGEAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERITONSILLAR ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA ESCHERICHIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONCUSSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEAR DROWNING (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD SODIUM INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PATELLOFEMORAL PAIN SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TORTICOLLIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OVARIAN ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CEREBRAL HYPOPERFUSION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONVULSION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PARKINSON'S DISEASE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
THALAMIC INFARCTION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENTAL DISORDER (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CYSTITIS GLANDULARIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY PARALYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHOSTASIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preladenant 2 mg (N=218) | Preladenant 5 mg (N=215) | Preladenant 5 mg (on Placebo in Parent Study) (N=106) | Preladenant 10 mg (N=96) | Rasagiline 1 mg (N=93) | Rasagiline 1 mg (on Placebo in Parent Study) (N=108)
CONSTIPATION (Gastrointestinal disorders) | 9 (10) | 12 (14) | 7 (7) | 5 (5) | 1 (1) | 3 (5)
NAUSEA (Gastrointestinal disorders) | 6 (6) | 8 (11) | 3 (3) | 1 (1) | 2 (2) | 7 (8)
FATIGUE (General disorders) | 7 (7) | 6 (6) | 3 (3) | 5 (5) | 0 (0) | 2 (2)
NASOPHARYNGITIS (Infections and infestations) | 12 (14) | 7 (7) | 3 (3) | 2 (2) | 4 (4) | 7 (7)
URINARY TRACT INFECTION (Infections and infestations) | 10 (10) | 10 (12) | 6 (7) | 5 (9) | 2 (2) | 6 (6)
FALL (Injury, poisoning and procedural complications) | 7 (8) | 16 (21) | 5 (5) | 3 (3) | 3 (3) | 4 (5)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 7 (7) | 4 (5) | 1 (1) | 5 (5) | 3 (3) | 1 (1)
WEIGHT DECREASED (Investigations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 5 (5) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3) | 0 (0) | 5 (7) | 2 (2) | 9 (10)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (7) | 7 (7) | 1 (1) | 3 (3) | 5 (6)
DYSKINESIA (Nervous system disorders) | 10 (11) | 19 (22) | 5 (6) | 8 (12) | 8 (8) | 9 (11)
PARKINSON'S DISEASE (Nervous system disorders) | 10 (12) | 12 (13) | 4 (5) | 4 (6) | 3 (3) | 0 (0)
TREMOR (Nervous system disorders) | 5 (5) | 2 (2) | 1 (1) | 5 (5) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early due to the lack of efficacy of preladenant in the parent studies NCT1155466 and NCT01227265.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the Sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication (including, without limitation, slides and texts of oral or other public presentations and texts of any transmission through any electronic media, eg, any computer access system such as the Internet, World Wide Web, etc) that report any results of the trial.